CLINICAL TRIAL: NCT03733470
Title: Pilot Study for Perfusion Heterogeneity: a Mechanistic Image-Based Emphysema Phenotype
Brief Title: Hypoxic Pulmonary Vasoconstriction Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eric A. Hoffman (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Eric A. Hoffman, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201101707; 5R01HL112986 (NIH)
Record Dates: First submitted 2018-10-23; First posted 2018-11-07 (Actual); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-08

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nonsusceptible Smokers (NS) (Experimental): 8 subjects recruited to study non-contrast imaging at TLC and 20%VC and with contrast using DECT to assess perfused blood volume. For the intervention, the subject will be administered 20 mg of Sildenafil and then the same scanning will be repeated one hour after sildenafil administration.
  Interventions: Drug: Sildenafil study group
- Susceptible Smokers (SS) (Experimental): 11 subjects recruited to study non-contrast imaging at TLC and 20% VC and with contrast using DECT to assess pefused blood volume. For the intervention the subject will be administered 20 mg of Sildenafil and then the same scanning will be repeated one hour after sildenafil administration.
  Interventions: Drug: Sildenafil study group

INTERVENTIONS:
Drug: Sildenafil study group — One dose of 20 mg Sildenafil will be given one hour before CT imaging.
  Other Names: Revatio

SUMMARY:
The purpose of this study is to determine if the events leading to smoking-associated centrilobular and paraseptal emphysema are caused by a failure of the lungs' inherent mechanisms to block hypoxic pulmonary vasoconstriction (HPV) in areas of smoking-induced inflammation.

DETAILED DESCRIPTION:
Overall goals of this study are to 1) determine the effects on sildenafil on the heterogeneity perfused blood volume in smokers susceptible to emphysema using dual energy CT 2) utilize pulmonary blood volume heterogeneity as an image-based biomarker to differentiate normal and susceptible smokers.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 30 and 60.
* Must be currently smoking at least 1/2 pack/day (confirmed with cotinine level).
* Must have pulmonary function test (PFT) results that meet the following:
* Forced Expiratory Volume at one second (FEV1)/Forced Vital Capacity (FVC) > 70%
* Forced Expiratory Flow at 25-75% (FEF25-75) > 79% of predicted
* FVC greater than 80% of predicted
* Must be able to give informed consent for self.

Exclusion Criteria:

* Pregnant or breastfeeding females.
* Body Mass Index (BMI) greater than 32.
* Weight of greater than 220 pounds (100 kg).
* Allergies to shell fish, seafood, eggs or iodine.
* Heart disease, kidney disease or diabetes.
* Diagnosis of asthma.
* Usage of any medications that are known to affect the heart or lungs (contraceptives, anti-depressants, analgesics EXCEPT aspirin, antihypertensives, and medications for osteoporosis and gastrointestinal diseases will be allowed).
* Any metal in or on the body between the nose and the abdomen.
* Any major organ system disease (by judgment of study medical team).

For the subjects that will receive Sildenafil as part of the study, additional exclusion criteria are as follows:

* Nitroglycerin usage.
* Prior history of hypersensitivity to Sildenafil.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-06-29 (Actual); Primary Completion 2014-01-13 (Actual); Study Completion 2014-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Hoffman, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
CT images will be shared including non-contrast images at Total Lung Capacity (TLC), Functional Residual Capacity (FRC) and Residual Volume (RV) as well as dual energy CT image data used to assess regional perfused blood volume. All associated pulmonary function test results will be shared. CT-derived metrics
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available starting 6 months after publication of the primary results of each aim.
Access Criteria: Data will be provided to academic-based researchers upon written request to the PI, Eric A. Hoffman, Ph.D. A nominal charge will be made for the time it takes for a technician to prepare and transfer the requested data. This costs will not exceed $250. This service will be available for a minimum of 2 years of study close.

REFERENCES:
- [Result] Alford SK, van Beek EJ, McLennan G, Hoffman EA. Heterogeneity of pulmonary perfusion as a mechanistic image-based phenotype in emphysema susceptible smokers. Proc Natl Acad Sci U S A. 2010 Apr 20;107(16):7485-90. doi: 10.1073/pnas.0913880107. Epub 2010 Apr 5. PMID 20368443
- Available data/document: Individual Participant Data Set: Data Distribution — http://www.i-clic.uihc.uiowa.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 22 subjects, 3 were eliminated because of blood pressure or asthma medications leaving 8NS and 11SS subjects.
Groups:
- Nonsusceptible Smokers (NS); Susceptible Smoker (SS): 22 subjects recruited. Pre-sildenafil we imaged with no contrast at TLC and 20% vital capacity (VC). To assess perfused blood volume (PBV), we imaged at 20% VC . For the intervention, the subject were administered 20 mg of oral Sildenafil and PBV imaging was repeated one hour after sildenafil.
  One group was labeled emphysema non-susceptible (NS) and another was emphysema susceptible (SS) based upon visual identification of emphysema in non-contrast CT scans. Of 22 subjects, 3 were eliminated because of blood pressure or asthma medications and two more were eliminated after scanning because of mis-matched pre and post sildenafil lung volumes, leaving 7NS and 10SS subjects. The study was designed to determine if the NS subjects have a greater coefficient of variation (CV) within 30x30x40 regions (approximately the size of an acinus) and whether sildenafil would eliminate the difference between medians of the per block CV histograms for NS and SS.
Period: Overall Study
Arm/Group | Nonsusceptible Smokers (NS) | Susceptible Smoker (SS)
Started | 8 | 11
Completed | 7 | 10
Not Completed | 1 | 1
Not completed — PI Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: 2 subjects were eliminated after scanning because of mis-matched pre and post sildenafil lung volumes, leaving 7NS and 10SS subjects.
Groups:
- Nonsusceptible Smokers (NS): 8 emphysema nonsusceptible smokers recruited to study non-contrast imaging at TLC and 20%VC and with contrast using DECT to assess perfused blood volume. For the intervention, the subject will be administered 20 mg of Sildenafil and then the same scanning will be repeated one hour after sildenafil administration.
- Susceptible Smokers (SS): 11 emphysema susceptible smokers recruited to study non-contrast imaging at TLC and 20%VC and with contrast using DECT to assess perfused blood volume. For the intervention, the subject will be administered 20 mg of Sildenafil and then the same scanning will be repeated one hour after sildenafil administration.
- Total: Total of all reporting groups
Arm/Group | Nonsusceptible Smokers (NS) | Susceptible Smokers (SS) | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 subjects were eliminated after scanning because of mis-matched pre and post sildenafil lung volumes, leaving 7NS and 10SS subjects
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 7 | 10 | 17
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 subjects were eliminated after scanning because of mis-matched pre and post sildenafil lung volumes, leaving 7NS and 10SS subjects.
  Participants
    Female | 6 | 9 | 15
    Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Perfused Blood Volume Assessed for a Change in Lung Inflammation Pre and Post Dose Sildenafil Administration
Description: Perfused blood volume will be measured by CT scan at two time points and compared at two points, pre and post the administration of sildenafil.
Time Frame: Change of perfused blood volume from baseline at one hour after sildenafil administration.
Measure: Mean (Standard Deviation); unit: coefficient of variation
Groups:
- Nonsusceptible Smokers (NS): 7 subjects recruited to study non-contrast imaging at TLC and 20%VC and with contrast using DECT to assess perfused blood volume. For the intervention, one dose of 20 mg Sildenafil was administered 20 mg of Sildenafil and then the same scanning will be repeated one hour after sildenafil administration.
  One dose of 20 mg Sildenafil will be given one hour before CT imaging.
- Susceptible Smoker (SS): 10 subjects recruited to study non-contrast imaging at TLC and 20%VC and with contrast using DECT to assess perfused blood volume. For the intervention, one dose of 20 mg Sildenafil was administered 20 mg of Sildenafil and then the same scanning will be repeated one hour after sildenafil administration.
  One dose of 20 mg Sildenafil will be given one hour before CT imaging.
Arm/Group | Nonsusceptible Smokers (NS) | Susceptible Smoker (SS)
Number analyzed (Participants) | 7 | 10
coefficient of variation | 0.37 (0.03) | 0.42 (0.09)
Statistical Analysis 1: Comparison: Nonsusceptible Smokers (NS) vs Susceptible Smoker (SS); Test type: Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Through study completion, one study visit.
Groups:
- Susceptible Smokers (SS): 11 subjects recruited to study non-contrast imaging at TLC and 20%VC and with contrast using DECT to assess perfused blood volume. For the intervention, the subject will be administered 20 mg of Sildenafil and then the same scanning will be repeated one hour after sildenafil administration.
Arm/Group | Nonsusceptible Smokers (NS) | Susceptible Smokers (SS)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/8 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No